CLINICAL TRIAL: NCT02582905
Title: Clinical Medication Development for Bipolar Disorder and Alcohol Use Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sherwood Brown, MD, PhD (Other)
Collaborators: University of Miami (Other); University of Texas Rio Grande Valley (Other)
Responsible Party: Sponsor-Investigator, Sherwood Brown, MD, PhD, Professor of Psychiatry, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 072014-005
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Alcohol Use Disorder; Bipolar Disorder; Schizoaffective Disorder Bipolar Type
Keywords: Alcohol Use Disorder; Bipolar Disorder; Mood; Alcohol craving; Pregnenolone; Citicoline
MeSH Terms: conditions — Alcoholism; Bipolar Disorder | interventions — Sugars; Cytidine Diphosphate Choline; Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo given beginning at 1 capsule twice daily (BID) increasing to 2 capsules BID at week 1, 3 capsules BID at week 2, and 4 capsules BID at weeks 3-12.
  Interventions: Drug: Placebo
- Citicoline (Experimental): Citicoline will be given beginning at 250 mg BID with an increase to 500 mg BID at week 1, 750 mg BID at week 2, and 1000 mg BID at weeks 3-12.
  Interventions: Dietary Supplement: Citicoline
- Pregnenolone (Experimental): Pregnenolone will be given beginning at 50 mg BID with an increase to 100 mg BID at week 1, 150 mg BID at week 2, and 250 mg BID at weeks 3-12.
  Interventions: Drug: Pregnenolone

INTERVENTIONS:
Drug: Placebo — Inactive ingredient matching the active comparators in appearance.
  Other Names: Sugar pill
  Arms: Placebo
Dietary Supplement: Citicoline — Citicoline is an over-the-counter nutritional supplement that is used for neuroprotective effects. It is a naturally occurring neurochemical in the human body.
  Other Names: CDP-Choline; cytidine diphosphate-choline
  Arms: Citicoline
Drug: Pregnenolone — Pregnenolone is a naturally occurring neurosteroid that is synthesized from cholesterol in the adrenal glands and also in the brain. Pregnenolone produces other neuroactive steroids.
  Other Names: pregn-5-en-3β-ol-20-one
  Arms: Pregnenolone

SUMMARY:
Preclinical and clinical data as well as mechanistic justification have been presented suggesting citicoline and pregnenolone are each promising treatments for alcohol use in BPD. Both appear to have favorable side effect profiles and no known drug-drug interactions. Thus, they have the potential to be safely used in a dual diagnosis population already taking other medications. A 12-week, randomized, double-blind, parallel-group, placebo-controlled adaptive design study of citicoline and pregnenolone is proposed in 199 persons with alcohol use disorder and bipolar I or II disorder or schizoaffective disorder (bipolar type). The primary aim will be to assess change in alcohol use. Biomarkers of alcohol use, alcohol craving, mood and cognition will also be assessed. Relationships between neurosteroid and choline levels and the outcome measures will be explored.

DETAILED DESCRIPTION:
A 12-week, randomized, double-blind, parallel-group, placebo-controlled adaptive, Drop The Loser (DTL) design clinical trial of citicoline and pregnenolone will be conducted in 199 outpatients with bipolar I or II disorder or schizoaffective disorder (bipolar type) and current alcohol use disorder. Potential participants will be identified and an appointment will be arranged. At this appointment, informed consent will be obtained, and assessment procedures, including a review of inclusion and exclusion criteria, will be performed.

A structured clinical interview for Diagnostic Statistical Manual (DSM-5), Structured Clinical Interview for Disorders (SCID) will be performed to establish the diagnoses of bipolar I or II disorder and alcohol use disorder. Recent alcohol use (and, if present, other substance use) will be assessed using the Timeline Followback (TLFB) method. Drinking severity and withdrawal symptoms will be assessed through a variety of measures (e.g., Clinical Institute Withdrawal Assessment of Alcohol Use-Revised (CIWA-Ar), Penn Alcohol Craving Scale (PACS), Short Index of Problems (SIP)). Length of problem alcohol use will be assessed by asking "When did alcohol first start causing you problems?" Blood will be drawn for laboratory analyses including a complete blood count (CBC) and Comprehensive Metabolic Panel (includes a liver panel with AST, ALT as well as lipids and electrolytes), and GGT and carbohydrate-deficient transferrin (CDT) will be added at baseline (week 0) and weeks 6 and 12. Cognition, including the domains of memory, decision making, impulsivity, attention, and executive functioning will also be assessed at baseline and week 12 using the World Health Organization/University of California at Los Angeles Auditory-Verbal Learning Test (WHO-UCLA AVLT), Trail Making Test (TMT), and the Golden Stroop Color Word Test. Women of childbearing potential will receive a urine pregnancy test at baseline, week 6, and week 12 and will be counseled about effective contraceptive methods. A psychiatrist (PI or Co-I) will assess participants at baseline and weekly follow-up visits and will participate in the informed consent process. The active medication or placebo capsules will be initiated at baseline and increased weekly in weeks 1, 2 and 3 to achieve the target doses for citicoline (2000 mg/day) or pregnenolone (500 mg/day). Side effects will be managed in a blinded fashion. Safety and side effects will be assessed with the Systematic Assessment for Treatment Emergent Events (SAFTEE). At weekly visits, mood and suicidality will be assessed through various measures (e.g. Hamilton Rating Scale for Depression (HRSD17), Columbia Suicide Severity Rating Scale (CSSRS) and assessment of alcohol use will again be evaluated. All participants will receive Medical Monitoring (MM) as a psychosocial platform. After study completion, participants will be provided standard psychiatric care until outside referral is arranged.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men and women age 18-70 years old with bipolar I or II disorder or schizoaffective disorder (bipolar type)
* English or Spanish speaking
* Current diagnosis of alcohol use disorder with at least moderate severity (DSM-5 terminology)
* Alcohol use of at least an average of 28 drinks a week if male or an average of 21 drinks per week if female and an average of 3 drinking days a week in the 28 days prior to intake
* Current mood stabilizer therapy (defined as lithium, lamotrigine, carbamazepine, oxcarbazepine or an atypical antipsychotic) with stable dose for ≥ 28 days prior to randomization or valproate/divalproex at a stable dose for ≥ 90 days (longer period due to data suggesting valproate may decrease alcohol use in BPD)
* Diagnosis of substance use disorder other than alcohol, caffeine or nicotine is allowed if 1) alcohol is the self-identified substance of choice and 2) severity of other substance use disorder is ≤ moderate

Exclusion Criteria:

* Mood disorders other than bipolar I or II disorders or schizoaffective disorder bipolar type (e.g. bipolar NOS, cyclothymic disorders, schizophrenia, schizoaffective disorder depressive type, or unipolar depression based on the SCID); other disorders (e.g. anxiety, will be allowed)
* Baseline HRSD17 or YMRS scores ≥ 35 to exclude those with very severe mood symptoms at baseline
* Evidence of clinically significant alcohol withdrawal symptoms defined as a CIWA-Ar score of ≥ 10
* Current (last 28 days) treatment with naltrexone, acamprosate, disulfiram, or topiramate as these may also decrease alcohol use
* Oral contraceptives and hormone replacement therapy. This exclusion is due to a possible interaction with pregnenolone.
* Women with hormone sensitive conditions such as breast cancer, uterine cancer, ovarian cancer, endometriosis, uterine fibroids. These persons are excluded because pregnenolone is converted to estrogens.
* Vulnerable populations (e.g. pregnant, nursing, cognitively impaired, incarcerated)
* High risk for suicide defined as > 1 attempt in past 12 months that required medical attention, any attempt in the past 3 months or current suicidal ideation with plan and intent such that outpatient care is precluded
* Intensive outpatient treatment (defined as ≥3 visits each week) for substance abuse (AA, NA meetings, or less intensive counseling at baseline will be allowed)
* Severe/unstable condition (e.g. cirrhosis, poorly controlled hypertension) or laboratory/physical exam findings consistent with serious illness (e.g. abnormal electrolytes) or AST or ALT >3 times normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas Rio Grande Valley, Edinburg, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Citicoline | Pregnenolone
Started | 29 | 30 | 37
Completed | 18 | 20 | 23
Not Completed | 11 | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Citicoline | Pregnenolone | Total
Number analyzed (Participants) | 29 | 30 | 37 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.00 (8.98) | 49.40 (10.07) | 47.35 (10.11) | 48.19 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 18 | 43
  Male | 17 | 17 | 19 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 26 | 32 | 81
  Not Hispanic or Latino | 5 | 3 | 5 | 13
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 15 | 13 | 40
  White | 16 | 15 | 21 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
YMRS [Mean (Standard Deviation); unit: units on a scale] — The Young Mania Rating Scale (YMRS) is an 11-item, observer-rated measure of manic symptoms. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. There are well described anchor points for each grade of severity. Higher scores indicate greater symptom severity. The range of possible scores is 0-60.
  units on a scale | 10.76 (8.23) | 10.20 (7.01) | 11.14 (7.33) | 10.73 (7.45)
HRSD [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Rating Scale - Depression (HRSD) is an observer-rated measure of depressive symptomatology. The individual item scores range from 0-4, 0-3 or 0-2 depending on the question. Higher scores indicate greater depressive symptom severity. The range of possible scores is 0-52.
  units on a scale | 14.62 (6.14) | 15.50 (7.13) | 13.46 (6.91) | 14.45 (6.74)
HRSA [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Rating Scale - Anxiety (HRSA) is a 14-item observer-rated assessment of anxiety. It consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Higher scores indicate greater anxiety symptom severity. The range of possible scores is 0-56.
  units on a scale | 13.07 (7.27) | 13.80 (6.67) | 14.19 (8.51) | 13.73 (7.54)
IDS-SR [Mean (Standard Deviation); unit: units on a scale] — The Inventory of Depressive Symptoms Self-Report (IDS-SR) is a 30-item self-report scale of depressive symptoms. Scores on each item range from 0-3. Higher scores indicate greater depressive symptom severity. The range of scores is 0-84.
  units on a scale | 26.00 (14.38) | 30.07 (16.57) | 26.92 (14.46) | 27.60 (15.05)
CIWA-Ar [Mean (Standard Deviation); unit: units on a scale] — The Clinical Institute of Withdrawal Assessment of Alcohol (CIWA-Ar) scale is a 10-item, clinician-rated scale of alcohol withdrawal symptoms. Each item scores range from 0-7. Higher scores indicate greater withdrawal symptom severity. The range of possible scores is 0-67.
  units on a scale | 3.64 (3.84) | 3.40 (2.85) | 2.97 (3.47) | 3.31 (3.38)
PACS [Mean (Standard Deviation); unit: units on a scale] — The Penn Alcohol Craving Scale (PACS) is a 5-item questionnaire that measures an individual's craving to drink alcohol in the past week. Each item scores range from 0-6. Higher scores indicate greater craving. The range of possibe score is 0-30.
  units on a scale | 19.72 (6.60) | 19.31 (7.90) | 17.65 (7.47) | 18.79 (7.33)
Metabolic Panel (AST) [Mean (Standard Deviation); unit: U/L] — A comprehensive metabolic panel (CMP) is a routine blood test that measures 14 different substances in a sample of blood. It provides information about one's metabolism and the balance of certain chemicals in the body. Aspartate aminotransferase (AST) is an enzyme typically found in the liver and is used to assess liver health. High AST values may indicate an underlying medical condition (e.g., liver condition).
  U/L | 23.82 (10.59) | 23.00 (8.39) | 24.38 (13.73) | 23.81 (11.35)
Metabolic Panel (ALT) [Mean (Standard Deviation); unit: U/L] — A comprehensive metabolic panel (CMP) is a routine blood test that measures 14 different substances in a sample of blood. It provides information about one's metabolism and the balance of certain chemicals in the body. Alanine transaminase (ALT) is an enzyme typically found in the liver and is used to assess liver health. High ALT values may indicate an underlying medical condition (e.g., liver condition).
  U/L | 22.96 (14.99) | 22.27 (9.15) | 24.51 (24.71) | 23.40 (18.33)
Metabolic Panel (GGT) [Mean (Standard Deviation); unit: U/L] — A comprehensive metabolic panel (CMP) is a routine blood test that measures 14 different substances in a sample of blood. It provides information about one's metabolism and the balance of certain chemicals in the body. Gamma-glutamyl transferase (GGT) is an enzyme typically found in the liver and is used to assess liver health. High GGT values may indicate an underlying medical condition (e.g., liver condition).
  U/L | 52.85 (73.46) | 36.50 (26.22) | 37.46 (27.07) | 41.80 (46.03)
Metabolic Panel (CDT) [Mean (Standard Deviation); unit: mg/L] — A comprehensive metabolic panel (CMP) is a routine blood test that measures 14 different substances in a sample of blood. It provides information about one's metabolism and the balance of certain chemicals in the body. Carbohydrate-deficient transferrin (CDT) is a blood plasma glycoprotein that carries iron through the blood to bone marrow. It is used as a biomarker of chronic alcohol intake. High CDT values indicate greater alcohol intake.
  mg/L | 57.39 (17.15) | 58.04 (27.06) | 58.72 (24.18) | 58.12 (22.97)
TLFB (Drinks per Drinking Day) [Mean (Standard Deviation); unit: Standard Drinks per Drinking Day] — The Timeline Follow Back (TLFB) - Alcohol is a clinician-completed assessment calendar that allows for an estimate of an individual's daily drinking habits over time (i.e., "prior 30 days" at baseline and "since last visit" during the study). Drinks per drinking day is calculated as the average number of standard drinks consumed, per each day indicated as a day during which alcohol was consumed, adjusted for the period of time being assessed (e.g., 30 days at baseline).
  Standard Drinks per Drinking Day | 9.15 (5.22) | 8.01 (3.61) | 7.35 (3.60) | 8.11 (4.17)

OUTCOME MEASURES:

1. Primary Outcome: Baseline-to-Exit Change in Drinks Per Drinking Day (TLFB)
Description: The Timeline Follow Back (TLFB) - Alcohol is a clinician-completed assessment calendar that allows for an estimate of an individual's daily drinking habits over time (i.e., "prior 30 days" at baseline and "since last visit" during the study). Drinks per drinking day is calculated as the average number of standard drinks consumed, per each day indicated as a day during which alcohol was consumed, adjusted for the period of time being assessed (e.g., 30 days at baseline). Baseline-to-Exit Change in Drinks per Drinking Day (TLFB) was calculated as Drinks/Drinking Day (Exit) - Drinks/Drinking Day (Baseline), with negative scores indicating a decrease in the number of drinks per drinking day. The TLFB (Timeline Followback) is a method of assessment of alcohol consumption and is not a scale with minimum and maximum values.
Time Frame: 12 weeks
Population: Participants having at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: Standard Drinks per Drinking Day
Arm/Group | Placebo | Citicoline | Pregnenolone
Number analyzed (Participants) | 29 | 30 | 37
Standard Drinks per Drinking Day | -1.98 (4.68) | -2.82 (3.84) | -1.22 (3.45)

2. Secondary Outcome: Examine the Use of an Adaptive Design in a Clinical Trial for Alcohol Use Disorder.
Description: A two-phase adaptive drop-the-loser (DTL) design was incorporated. A planned interim analysis was to be conducted after 50% of participants (n = 99) had been enrolled (phase 1), in which both treatments were to be compared to placebo. Predetermined decision rules were to be applied for dropping a treatment failing to show clinically meaningful efficacy over placebo: (1) The trial will be stopped if neither active treatment appears to be effective (Cohen's d < 0.25) and (2) The trial will continue to phase 2 (re-randomization) if there is evidence that at least one treatment is more effective than placebo. If both treatments were more effective, the trial was to continue with three arms.
Time Frame: Study Month 30
Population: Planned interim analyses were to be conducted after 50% of participants (n = 99) were enrolled (phase 1) to determine whether to proceed with a two-arm trial in phase 2 (i.e., drop-the-loser). Only upon proceeding to phase 2 could this aim be tested. Due to low enrollment (total enrolled: n=96), the required data necessary to test this aim was not obtained. As such, the study remained in phase 1 (with three arms), and the adaptive drop-the-loser design was untested.
Arm/Group | Placebo | Citicoline | Pregnenolone
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: Specific adverse events (AEs) and symptoms reported by more than one participant are grouped by the specific AE or symptom. Symptoms that were reported only once are grouped by system (e.g., respiratory, GI, etc.). AEs of participants who presented the same symptom during their follow-up visit were included only once in reporting.
Arm/Group | Placebo | Citicoline | Pregnenolone
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/37
Serious Adverse Events (participants affected / at risk) | 3/29 | 2/30 | 4/37
Other Adverse Events (participants affected / at risk) | 11/29 | 9/30 | 7/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | Citicoline (N=30) | Pregnenolone (N=37)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Admitted to hospital with panic attack
Suicide attempts (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) — Overdose and a psychiatric hospitalization
Inpatient alcohol treatment (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) — Three participants were admitted for inpatient alcohol treatment.
Overdose by partner on study medication (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — The partner of a participant overdosed on study medication.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — A participant was hospitalized with pneumonia.
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — A participant developed hyponatremia and was hospitalized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | Citicoline (N=30) | Pregnenolone (N=37)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea or vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Blurry vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Weight gain or increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Sedation (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Increased urinary frequency or difficulty (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Fractured bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3)
Numbness or tingling (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Decreased libido (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Cognitive difficulty (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Panic and anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Increased perspiration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Dental abscess (General disorders) | 0 (0) | 1 (1) | 0 (0)
Increased thirst (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Increased alcohol use (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Possible liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vivid dreams (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Metallic taste (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Motor vehicle accident (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 0 (0) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to low enrollment, the secondary aim (Examine the use of an adaptive design in a clinical trial for BPD and alcohol use disorder) was untested. Phase 1 of the adaptive design could not be completed as we were unable to enroll n = 99 participants. Therefore, we never reached the point of dropping a group and could not test the design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT02582905/Prot_SAP_000.pdf